CLINICAL TRIAL: NCT07333326
Title: Uterine Artery Doppler Flow Velocimetry Parameters for Predicting the Occurrence of Persistent Gestational Trophoblastic Neoplasia After Evacuation of Complete Hydatiform Mole ( a Prospective Cohort Study)
Brief Title: Uterine Artery Doppler Flow Velocimetry Parameters for Predicting the Occurrence of Persistent Gestational Trophoblastic Neoplasia After Evacuation of Complete Hydatiform Mole
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Montaser Ismail, Principal investigator, Minia University
Other Study IDs: UD-GTN-2025-1
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Gestational Trophoblastic Neoplasia; Complete Hydatiform Mole
Keywords: Gestational trophoblastic neoplasia
MeSH Terms: conditions — Gestational Trophoblastic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Prospective study will be conducted To copare uterine blood flow using Doppler ultrasound before and after evacuation of hydatiform mole between female patients with remissions and those with development of post-molar persistent gestational trophoblastic neoplasia to detect accuracy,efficacy,predictive value and acceptability of uterine artery doppler in predicting gestional trophoblastic neoplasia .

DETAILED DESCRIPTION:
Progression of complete hydatidiform mole to gestational trophoblastic neoplasia was reported to occur in 9 - 20% of patients. Suction curettage is considered the standard method of complete hydatiform mole evacuation .

Identification of occurrence of post-molar malignancy was detected during follow-up by serial assessment of serum human chorionic gonadotropin (hCG) . hCG rising or plateau mostly points to progression to malignancy thus requiring chemotherapy.Predicting liability to occurrence of post-molar malignancy mainly in patients with difficult continuous assessment of hCG is very important for adequate prompt management avoiding exposure to unnecessary chemotherapy .

There are many established predictive factors of post-molar malignancy as; patients age, size of ovaries, size of uterus, previous molar pregnancy, serial assessment of hCG level ,levels of vascular endothelial growth factor,TGF- beta 3 and HIF- 1alpha.

Moreover Trans-vaginal ultrasound with power Doppler might be used as a predictive factor for delayed response and resistance to chemotherapy particularly low-risk trophoblastic diseases .

Pelvic Doppler ultrasound is considered an essential diagnostic tool for evaluating uterine size and blood flow in patients with gestational trophoblastic neoplasia.

Additionally changes in flow resistance might be able to assess appropriate chemotherapeutic regimen for management of gestational trophoblastic neoplasia in addition to evaluating chemotherapy response .

Dopplerultrasound which is anoninvasive procedure for functional assessment of neo-vascularization,could assess patterns of highly abnormal flow in cases with invasive gestational trophoblastic neoplasia about two weeks post-evacuation before appearance of gross lesions and before marked risng hCG levels .

However, it is still controversial whether evaluation of Doppler flow velocimetry (DFV)parameters of uterine artery was a good predictorof gestational trophoblastic neoplasia after complete hydatiform mole evacuation .

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of complete hydatiform mole.
* Hemodynamically stable patient .
* No contraindication for anesthetic materials used for the evacuation .
* Acceptance of possible prolonged follow up , repeated uterine artery doppler ultrasound ,repeated HCG tests

Exclusion Criteria:

* Patient refusal to participate in the study.
* Patient with incomplete hydatiform mole .
* Patients who were lost during the follow-up period after this procedure.
* Contraindication for anesthetic materials used for the evacuation .

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Female 18:45 years with complete hydatiform mole
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Uterine artery Doppler flow velocimetry | We will perform DFV of uterine arteries on both sides at admission and 4 - 6 weeks after evacuation.
  First the patient will evaluate the urinary bladder Positioning of patient:supine position Amidsagittal section of uterus and cervical canal is obtained and the transducer is moved laterally untill the paracervical vessels are visualized color flow doppler is applied the uterine arteriesare seen as aliasing vessels along the side of the cervix Uterine artery doppler indices will be measured PSV=peak systolic velocity EDV=end diastolic velocity TAMV=time average medium velocity P.I(pulsatile index)=PSV-EDV/TAMV R.I(resistance index)=(PSV-EDV)/PSV SD(systolic diastolic ratio)=PSV/EDF

CONTACTS AND LOCATIONS:
Overall Officials: Montaser Ismail Mahmoud, Assistant lecturer, Principal Investigator — Minia University

IPD SHARING:
Plan to Share IPD: Undecided